CLINICAL TRIAL: NCT00168818
Title: A Phase III Randomised, Parallel Group, Double-blind, Active Controlled Study to Investigate the Efficacy and Safety of Two Different Dose Regimens of Orally Administered Dabigatran Etexilate Capsules [150 or 220 mg Once Daily Starting With Half Dose (75 or 110 mg) on the Day of Surgery] Compared to Subcutaneous Enoxaparin 40 mg Once Daily for 28-35 Days, in Prevention of Venous Thromboembolism in Patients With Primary Elective Total Hip Replacement Surgery. RE-NOVATE (Extended Thromboembolism Prevention After Hip Surgery)
Brief Title: Dabigatran Etexilate in Extended Venous Thromboembolism (VTE) Prevention After Hip Replacement Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1160.48; 2004-001988-21 (EudraCT Number: EudraCT)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2010-12-20 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-02

CONDITIONS: Thromboembolism; Arthroplasty, Replacement, Hip
MeSH Terms: conditions — Thromboembolism | interventions — Dabigatran; Enoxaparin

ARMS (3):
- dabigatran etexilate 75 mg (Experimental): daily dose 150 mg once daily, half a dose on the day of surgery
  Interventions: Drug: dabigatran etexilate
- dabigatran etexilate 110 mg (Experimental): daily dose 220 mg once daily, half a dose on the day of surgery
  Interventions: Drug: dabigatran etexilate
- enoxaparin (Active Comparator): 40 mg once daily
  Interventions: Drug: enoxaparin

INTERVENTIONS:
Drug: dabigatran etexilate — daily dose 150 mg once daily, half a dose on the day of surgery
  Arms: dabigatran etexilate 75 mg
Drug: dabigatran etexilate — daily dose 150 mg once daily, half a dose on the day of surgery
  Arms: dabigatran etexilate 110 mg
Drug: enoxaparin — 40 mg once daily
  Arms: enoxaparin

SUMMARY:
The objective of this study is to determine the comparative efficacy and safety of two oral regimens of dabigatran etexilate, compared to a standard subcutaneous regimen of enoxaparin, in prevention of venous thromboembolism in patients with primary elective total hip replacement surgery.

ELIGIBILITY:
Inclusion criteria

Inclusion criteria (selected):

* Patients (18 years or older) scheduled to undergo a primary, unilateral, elective total hip replacement
* Written Informed Consent

Exclusion criteria

Exclusion criteria (selected):

* Patients with an excessive risk of bleeding, for example because of history of bleeding diathesis major surgery or trauma within the last 3 months history of haemorrhagic stroke or any of the following intracranial pathologies: bleeding, neoplasm, AV malformation or aneurysm clinically relevant bleeding or gastric / duodenal ulcer within the last 6 months treatment with anticoagulants within 7 days prior to joint replacement surgery or anticipated need during the study treatment period thrombocytopenia.
* Active malignant disease or current cytostatic treatment
* Known severe renal insufficiency
* Liver disease expected to have any potential impact on survival, or elevated AST or ALT > 2x upper limit of normal
* Recent unstable cardiovascular disease or history of myocardial infarction within the last 3 months
* Pre-menopausal women who are pregnant or nursing, or are of child-bearing potential and are not practising or do not plan to continue practising acceptable methods of birth control
* Allergy to radio opaque contrast media or iodine, heparins (incl. heparin induced thrombocytopenia) or dabigatran
* Contraindications to enoxaparin
* Participation in a clinical trial during the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3494 (Actual)
Dates: Start 2004-11; Primary Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (116):
- Australia (10):
  - 1160.48.06108 Canberra Hospital, Garren, Australian Capital Territory
  - 1160.48.06106 St George Public Hospital, Kogarah, New South Wales
  - 1160.48.06110 Suite 13 level 4, Lismore, New South Wales
  - 1160.48.06105 Flinders Medical Centre, Bedford Park, South Australia
  - 1160.48.06104 Ecru, Box Hill, Victoria
  - 1160.48.06102 Monash Medical Centre, Clayton, Victoria
  - 1160.48.06101 Emeritus Research, Malvern, Victoria
  - 1160.48.06103 Maroondah Hospital, Ringwood East, Victoria
  - 1160.48.06113, Windsor, Victoria
  - 1160.48.06111 Haemophillia & Thrombosis Service, Perth, Western Australia
- Austria (4):
  - 1160.48.04304 Boehringer Ingelheim Investigational Site, Linz
  - 1160.48.04302 Boehringer Ingelheim Investigational Site, Vienna
  - 1160.48.04303 Boehringer Ingelheim Investigational Site, Wels
  - 1160.48.04301 Boehringer Ingelheim Investigational Site, Wiener Neustadt
- Belgium (7):
  - 1160.48.03207 UVC Brugmann, Brussels
  - 1160.48.03206 Campus Sint-Lucas, Ghent
  - 1160.48.03208 UZ Gent, Ghent
  - 1160.48.03202 Boehringer Ingelheim Investigational Site, Hasselt
  - 1160.48.03203 AZ Sint Elisabeth, Herentals
  - 1160.48.03205 Ziekenhuis Oost-Limburg, Lanaken
  - 1160.48.03201 UZ Gasthuisberg, Leuven
- Czechia (10):
  - 1160.48.42004 Boehringer Ingelheim Investigational Site, Brno-Bohunice
  - 1160.48.42010 Boehringer Ingelheim Investigational Site, Chomutov
  - 1160.48.42009 Boehringer Ingelheim Investigational Site, Havlíčkův Brod
  - 1160.48.42008 Boehringer Ingelheim Investigational Site, Jihlava
  - 1160.48.42002 Boehringer Ingelheim Investigational Site, Kladno
  - 1160.48.42006 Boehringer Ingelheim Investigational Site, Kolín
  - 1160.48.42003 Boehringer Ingelheim Investigational Site, Ostrava
  - 1160.48.42001 Boehringer Ingelheim Investigational Site, Pilsen
  - 1160.48.42007 Boehringer Ingelheim Investigational Site, Pradubice
  - 1160.48.42005 Boehringer Ingelheim Investigational Site, Prague
- Denmark (5):
  - 1160.48.04571 Boehringer Ingelheim Investigational Site, Hellerup
  - 1160.48.04570 Boehringer Ingelheim Investigational Site, Hørsholm
  - 1160.48.04573 Boehringer Ingelheim Investigational Site, København NV
  - 1160.48.04574 Boehringer Ingelheim Investigational Site, København S
  - 1160.48.04575 Boehringer Ingelheim Investigational Site, Silkeborg
- Finland (5):
  - 1160.48.35803 Boehringer Ingelheim Investigational Site, Helsinki
  - 1160.48.35802 Boehringer Ingelheim Investigational Site, Jyväskylä
  - 1160.48.35801 Boehringer Ingelheim Investigational Site, Oulu
  - 1160.48.35804 Boehringer Ingelheim Investigational Site, Seinäjoki
  - 1160.48.35805 Boehringer Ingelheim Investigational Site, Tampere
- France (4):
  - 1160.48.03304 Boehringer Ingelheim Investigational Site, Amiens
  - 1160.48.03303 Boehringer Ingelheim Investigational Site, Roubaix
  - 1160.48.03302 Boehringer Ingelheim Investigational Site, Soyaux
  - 1160.48.03308 Boehringer Ingelheim Investigational Site, Strasbourg
- Germany (11):
  - 1160.48.04906 Caritaskrankenhaus, Bad Mergentheim
  - 1160.48.04910 F.-A.-Universität Erlangen-Nürnberg, Erlangen
  - 1160.48.04904 Orthopädische Universitätsklinik, Frankfurt
  - 1160.48.04902 Klinikum Garmisch-Partenkirchen, Garmisch-Partenkirchen
  - 1160.48.04914 St. Bernhard-Hospital, Kamp-Lintfort
  - 1160.48.04907 Johannes Gutenberg-Universität Mainz, Mainz
  - 1160.48.04912 Orthopädische Klinik Markgröningen gGmbH, Markgröningen
  - 1160.48.04901 Kreiskrankenhaus, Rheinfelden
  - 1160.48.04915 Orthopädische Klinik Lindenlohe, Schwandorf in Bayern
  - 1160.48.04903 Hellmuth-Ulrici-Kliniken, Sommerfeld
  - 1160.48.04905 Aukammklinik, Wiesbaden
- Hungary (7):
  - 1160.48.03607 Boehringer Ingelheim Investigational Site, Békéscsaba
  - 1160.48.03603 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.48.03606 Boehringer Ingelheim Investigational Site, Budapest
  - 1160.48.03601 Boehringer Ingelheim Investigational Site, Gyula
  - 1160.48.03604 Boehringer Ingelheim Investigational Site, Kecskemét
  - 1160.48.03602 Boehringer Ingelheim Investigational Site, Szeged
  - 1160.48.03605 Boehringer Ingelheim Investigational Site, Székesfehérvár
- Italy (4):
  - 1160.48.03903 Boehringer Ingelheim Investigational Site, Bergamo
  - 1160.48.03904 Boehringer Ingelheim Investigational Site, Bologna
  - 1160.48.03902 Boehringer Ingelheim Investigational Site, Milan
  - 1160.48.03901 Boehringer Ingelheim Investigational Site, Pavia
- Netherlands (6):
  - 1160.48.03102 Boehringer Ingelheim Investigational Site, Amsterdam
  - 1160.48.03101 Boehringer Ingelheim Investigational Site, Heemstede
  - 1160.48.03107 Boehringer Ingelheim Investigational Site, Helmond
  - 1160.48.03103 Boehringer Ingelheim Investigational Site, Hilversum
  - 1160.48.03104 Boehringer Ingelheim Investigational Site, Nijmegen
  - 1160.48.03105 Boehringer Ingelheim Investigational Site, Sittard
- Norway (6):
  - 1160.48.04703 Boehringer Ingelheim Investigational Site, Ålesund
  - 1160.48.04701 Boehringer Ingelheim Investigational Site, Bodø
  - 1160.48.04704 Boehringer Ingelheim Investigational Site, Bærum Postterminal
  - 1160.48.04707 Boehringer Ingelheim Investigational Site, Bærum Postterminal
  - 1160.48.04706 Boehringer Ingelheim Investigational Site, Elverum
  - 1160.48.04702 Boehringer Ingelheim Investigational Site, Skien
- Poland (12):
  - 1160.48.04810 Boehringer Ingelheim Investigational Site, Bialystok
  - 1160.48.04804 Boehringer Ingelheim Investigational Site, Kielce
  - 1160.48.04806 Boehringer Ingelheim Investigational Site, Krakow
  - 1160.48.04807 Boehringer Ingelheim Investigational Site, Krakow
  - 1160.48.04812 Boehringer Ingelheim Investigational Site, Krakow
  - 1160.48.04820 Boehringer Ingelheim Investigational Site, Lodz
  - 1160.48.04814 Boehringer Ingelheim Investigational Site, Mielec
  - 1160.48.04808 Boehringer Ingelheim Investigational Site, Piekary Śląskie
  - 1160.48.04817 Boehringer Ingelheim Investigational Site, Rzeszów
  - 1160.48.04801 Boehringer Ingelheim Investigational Site, Warsaw
  - 1160.48.04802 Boehringer Ingelheim Investigational Site, Warsaw
  - 1160.48.04803 Boehringer Ingelheim Investigational Site, Warsaw
- South Africa (4):
  - 1160.48.02701 Boehringer Ingelheim Investigational Site, Bryanston
  - 1160.48.02704 Boehringer Ingelheim Investigational Site, Johannesburg
  - 1160.48.02703 Boehringer Ingelheim Investigational Site, Randburg
  - 1160.48.02702 Boehringer Ingelheim Investigational Site, Sandton
- Spain (11):
  - 1160.48.03405 Boehringer Ingelheim Investigational Site, Alcorcón (Madrid)
  - 1160.48.03403 Boehringer Ingelheim Investigational Site, Barcelona
  - 1160.48.03411 Boehringer Ingelheim Investigational Site, Barcelona
  - 1160.48.03407 Boehringer Ingelheim Investigational Site, Hospitalet (Barcelona)
  - 1160.48.03409 Boehringer Ingelheim Investigational Site, Jaén
  - 1160.48.03401 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.48.03402 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.48.03404 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.48.03406 Boehringer Ingelheim Investigational Site, Madrid
  - 1160.48.03408 Boehringer Ingelheim Investigational Site, Móstoles (Madrid)
  - 1160.48.03410 Boehringer Ingelheim Investigational Site, Valencia
- Sweden (10):
  - 1160.48.04602 Boehringer Ingelheim Investigational Site, Falköping
  - 1160.48.04601 Boehringer Ingelheim Investigational Site, Gothenburg
  - 1160.48.04607 Boehringer Ingelheim Investigational Site, Halmstad
  - 1160.48.04606 Boehringer Ingelheim Investigational Site, Kalmar
  - 1160.48.04603 Boehringer Ingelheim Investigational Site, Kungälv
  - 1160.48.04608 Boehringer Ingelheim Investigational Site, Lidköping
  - 1160.48.04605 Boehringer Ingelheim Investigational Site, Linköping
  - 1160.48.04604 Boehringer Ingelheim Investigational Site, Mölndal
  - 1160.48.04610 Boehringer Ingelheim Investigational Site, Stockholm
  - 1160.48.04609 Boehringer Ingelheim Investigational Site, Varberg

REFERENCES:
- [Derived] Eriksson BI, Dahl OE, Rosencher N, Clemens A, Hantel S, Feuring M, Kreuzer J, Huo M, Friedman RJ. Oral dabigatran etexilate versus enoxaparin for venous thromboembolism prevention after total hip arthroplasty: pooled analysis of two phase 3 randomized trials. Thromb J. 2015 Nov 17;13:36. doi: 10.1186/s12959-015-0067-8. eCollection 2015. PMID 26578849
- [Derived] Eriksson BI, Dahl OE, Rosencher N, Clemens A, Hantel S, Kurth AA. Efficacy of delayed thromboprophylaxis with dabigatran: pooled analysis. Thromb Res. 2012 Dec;130(6):871-6. doi: 10.1016/j.thromres.2012.08.315. Epub 2012 Sep 17. PMID 22995531
- [Derived] Rosencher N, Noack H, Feuring M, Clemens A, Friedman RJ, Eriksson BI. Type of anaesthesia and the safety and efficacy of thromboprophylaxis with enoxaparin or dabigatran etexilate in major orthopaedic surgery: pooled analysis of three randomized controlled trials. Thromb J. 2012 Jun 18;10(1):9. doi: 10.1186/1477-9560-10-9. PMID 22709460
- [Derived] Eriksson BI, Dahl OE, Rosencher N, Kurth AA, van Dijk CN, Frostick SP, Prins MH, Hettiarachchi R, Hantel S, Schnee J, Buller HR; RE-NOVATE Study Group. Dabigatran etexilate versus enoxaparin for prevention of venous thromboembolism after total hip replacement: a randomised, double-blind, non-inferiority trial. Lancet. 2007 Sep 15;370(9591):949-56. doi: 10.1016/S0140-6736(07)61445-7. PMID 17869635

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The treatment period is from first administration of study medication, until 3 days after last administration of study medication. Treatment duration is planned for 28 - 35 days. The study period is from first administration of study medication until day 84 - 91.
Pre-assignment Details: Whilst 3494 patients were enrolled/randomised to treatment prior to surgery in this trial, only 3463 started treatment. Therefore, 31 patients were randomised but not treated (treatment was planned to start post surgery).
Groups:
- Dabigatran 220mg: Patients were treated with 220mg dabigatran etexilate once daily as capsules for oral administration and placebo subcutaneous injections. Placebo injections matching the enoxaparin syringes.
- Dabigatran 150mg: Patients were treated with 150mg dabigatran etexilate once daily as capsules for oral administration and placebo subcutaneous injections. Placebo injections matching the enoxaparin syringes.
- Enoxaparin: Patients were treated with 40mg Enoxaparin once daily for subcutaneous injection and placebo capsules. Placebo capsules matching the dabigatran capsules.
Period: Overall Study
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Started | 1146 | 1163 | 1154
Completed | 1029 | 1054 | 1030
Not Completed | 117 | 109 | 124
Not completed — Adverse Event | 23 | 29 | 31
Not completed — Protocol Violation | 16 | 11 | 11
Not completed — Lost to Follow-up | 13 | 4 | 15
Not completed — Withdrawal by Subject | 43 | 41 | 37
Not completed — Other | 22 | 24 | 30
Period: Treatment
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Started | 1146 | 1163 | 1154
Completed | 1013 | 1012 | 1021
Not Completed | 133 | 151 | 133
Not completed — Adverse Event | 77 | 89 | 68
Not completed — Protocol Violation | 8 | 11 | 11
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Withdrawal by Subject | 25 | 20 | 22
Not completed — Other | 23 | 29 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin | Total
Number analyzed (Participants) | 1146 | 1163 | 1154 | 3463
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (10.4) | 63.4 (11.1) | 63.8 (10.8) | 63.9 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 636 | 667 | 651 | 1954
  Male | 510 | 496 | 503 | 1509
Body Mass Index N=(1146;1163;1151;3460) [Mean (Standard Deviation); unit: kg/m^2] | 27.7 (4.6) | 27.8 (4.6) | 27.5 (4.3) | 27.7 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Total Venous Thromboembolic Event and All-cause Mortality During Treatment Period
Description: Total Venous Thromboembolic Event (VTE) includes both proximal and distal deep vein thrombosis (DVT) (detected by routine bilateral venography), symptomatic DVT (confirmed by venous compression ultrasound, venography or autopsy) and pulmonary embolism (PE) (confirmed by pulmonary V-Q scintigraphy, chest x-ray, pulmonary angiography, spiral CT or autopsy).
  All of these components and all deaths were centrally adjudicated by the VTE events committee, which was not aware of the treatment allocation of the patients.
Time Frame: First administration until 31-38 days
Population: Full Analysis Set (all patients who had surgery and were randomised, received treatment, had an evaluable venogram for distal and proximal Deep Vein Thrombosis, or symptomatic Deep Vein Thrombosis, Pulmonary Embolism, or had died)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 880 | 874 | 897
Participants | 53 | 75 | 60
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Non-Inferiority or Equivalence — Non-inferiority Analysis with NI margin 7.7%. This results from the null-hypotheses of non-inferiority testing, where the rate difference has to be below 7.7%. Non-inferiority can only be shown with CI; p = 0.5648, Normal approximation — p-value is for superiority testing; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = -0.7, 95% CI [-2.9 to 1.6]
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.1339, Normal approximation — p-value is for superiority testing; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = 1.9, 95% CI [-0.6 to 4.4]

2. Secondary Outcome: Major Venous Thromboembolic Event and Venous Thromboembolic Event-related Mortality During Treatment Period
Description: Major Venous Thromboembolic Event (VTE) is defined as proximal DVT and PE, as adjudicated by the VTE events committee
Time Frame: First administration until 31-38 days
Population: Full Analysis Set - major (all patients who had surgery and were randomised, received treatment, had an evaluable venogram for proximal Deep Vein Thrombosis, or had confirmed symptomatic Deep Vein Thrombosis, Pulmonary Embolism, or had died by a Venous Thromboembolic Event-related death)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 909 | 888 | 917
Participants | 28 | 38 | 36
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.3256, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = -0.8, 95% CI [-2.5 to 0.8]
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.7052, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = 0.4, 95% CI [-1.5 to 2.2]

3. Secondary Outcome: Proximal Deep Vein Thrombosis During Treatment Period
Description: Proximal Deep Vein Thrombosis as adjudicated by the VTE events committee
Time Frame: First administration until 31-38 days
Population: Full Analysis Set - pDVT (all patients who had surgery and were randomised, received treatment, had an evaluable venogram for proximal Deep Vein Thrombosis, or had confirmed symptomatic Deep Vein Thrombosis)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 905 | 885 | 914
Participants | 23 | 35 | 33
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.1863, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = -1.1, 95% CI [-2.7 to 0.5]
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.7020, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = 0.3, 95% CI [-1.4 to 2.1]

4. Secondary Outcome: Total Deep Vein Thrombosis During Treatment Period
Description: Total Deep Vein Thrombosis as adjudicated by the VTE events committee
Time Frame: First administration until 31-38 days
Population: Full Analysis Set - tDVT (all patients who had surgery and were randomised, received treatment, had an evaluable venogram, or had confirmed symptomatic Deep Vein Thrombosis)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 874 | 871 | 894
Participants | 46 | 72 | 57
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.3173, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = -1.1, 95% CI [-3.3 to 1.1]
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Risk difference versus Enoxaparin; Test type: Superiority or Other; p = 0.1274, Normal approximation; Normal approximation of independent binomial distribution without stratification; Risk Difference (Percentage) = 1.9, 95% CI [-0.5 to 4.3]

5. Secondary Outcome: Symptomatic Deep Vein Thrombosis During Treatment Period
Description: Symptomatic Deep Vein Thrombosis, confirmed by venous compression ultrasound, venography or autopsy, and as adjudicated by the VTE events committee
Time Frame: First administration until 31-38 days
Population: Full Analysis Set - op (all patients who are treated and operated)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 1137 | 1156 | 1142
Participants | 6 | 9 | 1
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.0694, Fisher Exact
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.0212, Fisher Exact

6. Secondary Outcome: Pulmonary Embolism During Treatment Period
Description: Pulmonary embolism confirmed by pulmonary V-Q scintigraphy, chest x-ray, pulmonary angiography, spiral CT or autopsy, and as adjudicated by the VTE events committee
Time Frame: First administration until 31-38 days
Population: Full Analysis Set - op (all patients who are treated and operated)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 1137 | 1156 | 1142
Participants | 5 | 1 | 3
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.5062, Fisher Exact
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.3717, Fisher Exact

7. Secondary Outcome: Death During Treatment Period
Description: All cause death, as adjudicated by the VTE events committee
Time Frame: First administration until 31-38 days
Population: Full Analysis Set - op (all patients who are treated and operated)
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 1137 | 1156 | 1142
Participants | 3 | 3 | 0
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.1240, Fisher Exact
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.2497, Fisher Exact

8. Secondary Outcome: Total Venous Thromboembolic Event (VTE) and All-cause Mortality During the Follow-up Period
Description: Total Venous Thromboembolic Event (VTE) includes both proximal and distal deep vein thrombosis (DVT) (detected by routine bilateral venography), symptomatic DVT (confirmed by venous compression ultrasound, venography or autopsy) and pulmonary embolism (PE) (confirmed by pulmonary V-Q scintigraphy, chest x-ray, pulmonary angiography, spiral CT or autopsy).
Time Frame: end of treatment to day 91±7
Population: Patients with any data available during follow-up
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 1106 | 1117 | 1108
Participants
  Total VTE and all-cause mortality | 1 | 4 | 5
  asymptotic Deep Vein Thrombosis | 0 | 1 | 3
  symptotic Deep Vein Thrombosis | 1 | 1 | 0
  Pulmonary Embolism | 0 | 0 | 1
  death | 0 | 2 | 1

9. Secondary Outcome: Number of Participants With Bleeding Events (Defined According to Modified McMaster Criteria) During Treatment Period
Description: Major bleeding events were defined as
  * fatal
  * clinically overt associated with loss of haemoglobin >=20g/L in excess of what was expected
  * clinically overt leading to the transfusion of >=2 units packed cells or whole blood in excess of what was expected
  * symptomatic retroperitoneal, intracranial, intraocular or intraspinal
  * requiring treatment cessation
  * leading to re-operation
  Clinically-relevant was defined as
  * spontaneous skin hematoma greater than or equal to 25 cm²
  * wound hematoma greater than or equal to 100 cm²
  * spontaneous nose bleed lasting longer than 5 min
  * macroscopic hematuria spontaneous or lasting longer than 24 hours if associated with an intervention
  * spontaneous rectal bleeding (more than a spot on toilet paper)
  * gingival bleeding lasting longer than 5 min
  * any other bleeding event considered clinically relevant by the investigator
  Minor bleeding events were defined as all other bleeding events that did not fulfil the criteria from above.
Time Frame: First administration until 31-38 days
Population: Treated set
Measure: Number; unit: Participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 1146 | 1163 | 1154
Participants
  Major | 23 | 15 | 18
  Clinical relevant | 48 | 55 | 40
  Minor | 70 | 72 | 74
  None | 1005 | 1021 | 1022
Statistical Analysis 1: Comparison: Dabigatran 220mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.4352, Fisher Exact
Statistical Analysis 2: Comparison: Dabigatran 150mg vs Enoxaparin; Comparison versus Enoxaparin; Test type: Superiority or Other; p = 0.6037, Fisher Exact

10. Secondary Outcome: Blood Transfusion
Description: Blood transfusion for treated and operated patients on Day of surgery.
Time Frame: Day 1
Measure: Number; unit: participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 1137 | 1156 | 1142
participants
  Patients with >=1 transfusions | 517 | 531 | 542
  Patients with >=1 non-autologous transfusions | 259 | 266 | 286

11. Secondary Outcome: Volume of Blood Loss
Description: Volume of blood loss for treated and operated patients during surgery.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 1127 | 1147 | 1133
mL | 457 (304) | 435 (271) | 463 (291)

12. Secondary Outcome: Laboratory Analyses
Description: Frequency of patients with possible clinically significant abnormalities.
Time Frame: First administration to end of study
Population: Treated patients
Measure: Number; unit: participants
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Number analyzed (Participants) | 1103 | 1098 | 1103
participants
  AST increase N=(1103;1097;1103) | 11 | 16 | 29
  AST decrease N=(1103;1097;1103) | 0 | 0 | 0
  ALT increase N=(1103;1098;1103) | 28 | 29 | 59
  ALT decrease N=(1103;1098;1103) | 0 | 0 | 0
  Bilirubin increase N=(1102;1094;1102) | 25 | 24 | 34
  Bilirubin decrease N=(1102;1094;1102) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 13 weeks
Description: Treatment emergent events (last medication + 3 days)
Arm/Group | Dabigatran 220mg | Dabigatran 150mg | Enoxaparin
Serious Adverse Events (participants affected / at risk) | 89/1146 | 91/1163 | 82/1154
Other Adverse Events (participants affected / at risk) | 620/1146 | 642/1163 | 648/1154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran 220mg (N=1146) | Dabigatran 150mg (N=1163) | Enoxaparin (N=1154)
Acute myocardial infarction (Cardiac disorders) | 0 | 2 | 0
Acute right ventricular failure (Cardiac disorders) | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 3
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 3 | 5
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1
Angle closure glaucoma (Eye disorders) | 0 | 1 | 0
Diplopia (Eye disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 2
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 1
Drug ineffective (General disorders) | 2 | 1 | 0
Feeling hot and cold (General disorders) | 0 | 0 | 1
Impaired healing (General disorders) | 1 | 4 | 0
Inflammation of wound (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 3 | 2 | 0
Pyrexia (General disorders) | 2 | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1
Wound necrosis (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 0 | 2
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 0 | 0
Perineal abscess (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 1
Postoperative infection (Infections and infestations) | 1 | 0 | 1
Postoperative wound infection (Infections and infestations) | 4 | 2 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 3 | 0 | 2
Wound abscess (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 7 | 3 | 7
Wound infection staphylococcal (Infections and infestations) | 0 | 0 | 1
Arterial injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Bone fissure (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Device breakage (Injury, poisoning and procedural complications) | 1 | 0 | 2
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 3 | 6 | 6
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1 | 2
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 5 | 4 | 4
Joint dislocation postoperative (Injury, poisoning and procedural complications) | 0 | 0 | 2
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Operative haemorrhage (Injury, poisoning and procedural complications) | 2 | 0 | 3
Post procedural discharge (Injury, poisoning and procedural complications) | 1 | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 1
Postoperative thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 2
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 2
Wound secretion (Injury, poisoning and procedural complications) | 8 | 8 | 3
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 2
Oxygen saturation decreased (Investigations) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Langerhans' cell granulomatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 2 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Neurogenic bladder (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Prostatism (Reproductive system and breast disorders) | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 2
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Immobile (Social circumstances) | 1 | 0 | 0
Immobilisation prolonged (Social circumstances) | 1 | 0 | 0
Air embolism (Vascular disorders) | 0 | 1 | 0
Arterial rupture (Vascular disorders) | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 6 | 13 | 9
Haematoma (Vascular disorders) | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 2
Peripheral embolism (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 1 | 0
Wound haemorrhage (Vascular disorders) | 2 | 3 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabigatran 220mg (N=1146) | Dabigatran 150mg (N=1163) | Enoxaparin (N=1154)
Constipation (Gastrointestinal disorders) | 146 | 140 | 149
Nausea (Gastrointestinal disorders) | 238 | 258 | 289
Vomiting (Gastrointestinal disorders) | 193 | 185 | 191
Oedema peripheral (General disorders) | 62 | 79 | 56
Pyrexia (General disorders) | 121 | 140 | 162
Wound secretion (Injury, poisoning and procedural complications) | 94 | 88 | 60
Insomnia (Psychiatric disorders) | 77 | 88 | 80
Hypotension (Vascular disorders) | 81 | 76 | 81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract